CLINICAL TRIAL: NCT03849521
Title: In Vivo Atherosclerotic Plaque Calcium Characterization for Predicting Ruptured Plaques
Brief Title: Plaque Calcium Characterization and Ruptured Plaques
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Li Min (Other)
Responsible Party: Sponsor-Investigator, Li Min, Vice Director, Jinan Military General Hospital
Organization: Jinan Military General Hospital (Other)
Other Study IDs: 201703
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Vulnerable Atherosclerotic Plaque
Keywords: Atherosclerosis; Calcium; MR
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — The carotid plaques of patient undergoing carotid endarterectomy will be retented. Furthermore, the histopathological features as well as bone-like genetic program will be analyzed systematically.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asymptomatic group: Group with asymptomatic patients with carotid atherosclerosis.
  Interventions: Diagnostic Test: MRI
- Symptomatic group: Group with symptomatic patients with carotid atherosclerosis.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Enhanced carotid calcification presented by UTE MR.

SUMMARY:
Recently, ultrashort echo time (UTE) MR, which allows detection of the ultrashort T2 components, has been used to image plaque calcification in ex vivo carotid and coronary arteries. The results demonstrated that UTE images are able to identify plaque calcification and enables accurate quantification of calcium volumes. However, gadolinium-based contrast agents during in vivo CMR could not be performed in these ex vivo study. Agnese et al. believed that calcifications with 18F-NaF PET uptake might be considered to represent dormant areas where on-going mineralization, which is a key sign to identify and localise ruptured and high risk coronary plaque. We, therefore, hypothesize that enhanced carotid calcification presented by UTE MR may be a critical sign for symptomatic patients.

In this study, we will investigate the feasibility of enhanced UTE MR in human carotid arteries in vivo. Furthermore, we analyzed the correlation between UTE MR and microcalcification of in the carotid plaques. Based on the diagnostic ability of enhanced UTE MR for microcalcification, we will investigate the potential of enhanced calcification to distinguish symptomatic from asymptomatic patients with carotid atherosclerosis and research the prognostic ability of enhance calcufication in UTE MR.

DETAILED DESCRIPTION:
Atherosclerosis, characterized by the accumulation of lipids and inflammatory cells in the large arteries, is one of the most common causes of morbidity and mortality in developed and developing countries. Atherosclerotic plaque rupture-induced thrombosis or obstruction of artery is the most important cause for the sudden and unpredictable onset of acute artery stroke. Our understanding of specific characteristics of the vulnerable atherosclerotic plaque has been enhanced by retrospective pathological studies, which have identified common phenotypic features of the atherosclerotic plaque most prone to rupture and trigger thrombotic events. A thin fibrous cap, a large lipid core, high macrophage count, and intraplaque hemorrhage have all been identified as markers of the so-called "vulnerable" plaque being related to a higher stroke risk.

Calcification of atherosclerotic lesions was long thought to be an age - related, passive process where a combination of high local concentrations of phosphates and phosphatidylserines from necrotic cells and an absence of calcification inhibitors results in the precipitation of calcium phosphate particles. Recently increasingly data has revealed that atherosclerotic calcification is a more active process, involving complex signaling pathways and bone-like genetic programs. The distinction of early or active calcification as a destabilizing process and late calcification as a more stable state has also been supported by histological studies. This has lead to interest in characterizing early stages of calcification metabolically by making use of the positron emission tomography (PET)/CT imaging of atherosclerosis using 18F-sodium fluoride (18F-NaF), which has recently been reported having the potential to distinguish dormant areas with on-going mineralization and quiescent atherosclerotic calcium. Nevertheless, PET/CT is an expensive and a radioactive examination, which is not appropriate for large-scale screening or serial follow-up studies.

MRI is ideal for serial studies of lesions of atherosclerosis over time because it is noninvasive and is superior to other imaging modalities in distinguishing soft tissue contrast. In conventional gradient echo based MRI with TEs in the 1 to 2 ms range, however, the very short T2 relaxation time of solid calcifications on the order of some μs causes almost complete signal cancellation, which may cause significant overestimation of the calcified region and could not provide information about calcium density. Moreover, the low or zero signal from calcium with short T2 means that there is little opportunity to manipulate conspicuity by using different pulse sequences or contrast agents.

Recently, ultrashort echo time (UTE) MR, which allows detection of the ultrashort T2 components, has been used to image plaque calcification in ex vivo carotid and coronary arteries. The results demonstrated that UTE images are able to identify plaque calcification and enables accurate quantification of calcium volumes. However, gadolinium-based contrast agents during in vivo CMR could not be performed in these ex vivo study. Agnese et al. believed that calcifications with 18F-NaF PET uptake might be considered to represent dormant areas where on-going mineralization, which is a key sign to identify and localise ruptured and high risk coronary plaque. We, therefore, hypothesize that enhanced carotid calcification presented by UTE MR may be a critical sign for symptomatic patients.

In this study, we will investigate the feasibility of enhanced UTE MR in human carotid arteries in vivo. Furthermore, we analyzed the correlation between UTE MR and microcalcification of in the carotid plaques. Based on the diagnostic ability of enhanced UTE MR for microcalcification, we will investigate the potential of enhanced calcification to distinguish symptomatic from asymptomatic patients with carotid atherosclerosis and research the prognostic ability of enhance calcufication in UTE MR.

ELIGIBILITY:
Inclusion Criteria:

Patients referred for carotid endarterectomy or stent were prospectively enrolled.

Exclusion Criteria:

Patients with ferromagnetic metal, active implants such as pacemakers, aneurysm clips, known claustrophobia, and those who were unable to provide informed consent were excluded from enrollment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sixty patients referred for carotid endarterectomy or stent were prospectively enrolled.Patients gave written informed consent to participate in this Institutional Review Board-approved human subjects investigation. Clinical assessment at baseline using both patient interview and chart review documented presence or absence of symptoms (symptomatic and asymptomatic patients, respectively) attributable to the carotid artery disease, such as transient ischemic attack or cerebrovascular accident in the distribution of the diseased artery and absence of other source of embolism.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms attributable to the carotid artery disease | 3 years
  Clinical assessment at baseline using both patient interview and chart review documented presence or absence of symptoms (symptomatic and asymptomatic patients, respectively) attributable to the carotid artery disease, such as transient ischemic attack or cerebrovascular accident in the distribution of the diseased artery and absence of other source of embolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Min Li, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No